CLINICAL TRIAL: NCT00007644
Title: CSP #407 - Prostate Cancer Intervention Versus Observation Trial (PIVOT): A Randomized Trial Comparing Radical Prostatectomy Versus Palliative Expectant Management for the Treatment of Clinically Localized Prostate Cancer
Brief Title: Prostate Cancer Intervention Versus Observation Trial (PIVOT)
Acronym: PIVOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 407; NCT00002606 (obsolete NCT alias)
Record Dates: First submitted 2000-12-29; First posted 2001-01-01 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer
Keywords: cancer of the prostate (CAP); cancer treatment; chronic diseases; expectant management; genitourinary; prostate; prostate specific cancer mortality; radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radical Prostatectomy (Other): Surgical removal of the prostate
  Interventions: Procedure: Radical prostatectomy
- Watchful Waiting (No Intervention): Closely watching, waiting and treating symptoms if and when cancer progresses

INTERVENTIONS:
Procedure: Radical prostatectomy — Surgical removal of the prostate
  Arms: Radical Prostatectomy

SUMMARY:
Radical prostatectomy provides potentially curative removal of the cancer. However, it subjects patients to the morbidity and mortality of the surgery and may be neither necessary nor effective. Expectant management does not offer potential cure. However, it provides palliative therapy for symptomatic or metastatic disease progression, avoids potentially excessive and morbid interventions in asymptomatic patients, and emphasizes management approaches for focus on relieving symptoms while minimizing therapeutic complications.

The primary objective of this study is to determine which of two strategies is superior for the management of clinically localized CAP: 1) radical prostatectomy with early aggressive intervention for disease persistence or recurrence, 2) expectant management with reservation of therapy for palliative treatment of symptomatic or metastatic disease progression. Outcomes include total mortality, CAP mortality, disease free and progression free survival, morbidity, quality of life, and cost effectiveness.

DETAILED DESCRIPTION:
Primary Hypothesis: To determine whether radical prostatectomy or expectant management is more effective in reducing mortality and extending life.

Secondary Hypothesis: To determine which treatment strategy is superior in terms of prostate specific cancer mortality, quality of life, occurrence or recurrence of symptoms and need for cancer treatment.

Intervention: 1) Radical prostatectomy, plus intervention for evidence of disease persistence or recurrence, 2) Expectant management with palliative therapy reserved for symptomatic or metastatic disease progression.

Primary Outcomes: All cause mortality.

Study Abstract: Cancer of the prostate (CAP) is the most common nondermatologic and the second most frequent cause of cancer deaths in men. No cure is currently possible for disseminated disease. Cancer confined to the prostate is believed to be curable, with the most frequently recommended therapy being surgical extirpation of the tumor with radical prostatectomy. However, despite increasing cancer detection and aggressive surgical treatment, population-based mortality rates from prostate cancer have not decreased, neither nationally nor in states with high rates of radical prostatectomy. Existing evidence does not demonstrate the superiority of this procedure compared to expectant management in the treatment of localized prostate cancer. Data from case series suggest that either treatment approach provides equivalent all-cause as well as prostate cancer specific mortality. The only randomized trial was limited by a small sample size but the results favored expectant management.

Radical prostatectomy provides potentially curative removal of the cancer. However, it subjects patients to the morbidity and mortality of the surgery and may be neither necessary nor effective. Expectant management does not offer potential cure. However, it provides palliative therapy for symptomatic or metastatic disease progression, avoids potentially excessive and morbid interventions in asymptomatic patients, and emphasizes management approaches for focus on relieving symptoms while minimizing therapeutic complications.

The primary objective of this study is to determine which of two strategies is superior for the management of clinically localized CAP: 1) radical prostatectomy with early aggressive intervention for disease persistence or recurrence, 2) expectant management with reservation of therapy for palliative treatment of symptomatic or metastatic disease progression. Outcomes include total mortality, CAP mortality, disease free and progression free survival, morbidity, quality of life, and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically localized CAP
* Diagnosis of Prostate Cancer within previous 6 months
* Age 75 years or younger

Exclusion Criteria:

PSA > 50 ng/ml Bone scan consistent with metastatic disease Other evidence that cancer of the prostate is not clinically localized Diagnosis of prostate cancer greater than 12 months ago Life expectancy less than 10 years Serum creatinine greater than 3 mg/dl Myocardial infarction within last 6 months Unstable angina New York Heart Association Class III or IV congestive heart failure Severe pulmonary disease Lifer failure Severe dementia Debilitating illness Malignancies, except for nonmelanomatous skin cancer, in the last 5 years

Max Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 1994-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J. Wilt, MD MPH, Study Chair — Minneapolis Veterans Affairs Medical Center
Locations (31):
- United States (31):
  - VA Medical Center, Birmingham, Birmingham, Alabama
  - Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock, North Little Rock, Arkansas
  - VA Medical Center, Long Beach, Long Beach, California
  - VA Medical Center, San Francisco, San Francisco, California
  - VA Greater Los Angeles HCS, Sepulveda, Sepulveda, California
  - James A. Haley Veterans Hospital, Tampa, Tampa, Florida
  - VA Medical Center, Boise, Boise, Idaho
  - Jesse Brown VAMC (WestSide Division), Chicago, Illinois
  - Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana
  - VA Medical Center, Iowa City, Iowa City, Iowa
  - VA Medical Center, Lexington, Lexington, Kentucky
  - Overton Brooks VA Medical Center, Shreveport, Shreveport, Louisiana
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - VA New Jersey Health Care System, East Orange, East Orange, New Jersey
  - VA Stratton Medical Center, Albany, Albany, New York
  - New York Harbor Health Care System, Brooklyn, Brooklyn, New York
  - VA Western New York Healthcare System at Buffalo, Buffalo, New York
  - VA Medical Center, Syracuse, Syracuse, New York
  - VA Medical Center, Bronx, The Bronx, New York
  - VA Medical Center, Oklahoma City, Oklahoma City, Oklahoma
  - VA Medical Center, Portland, Portland, Oregon
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania
  - VA Medical Center, Providence, Providence, Rhode Island
  - VA Medical Center, Memphis, Memphis, Tennessee
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - Central Texas Veterans Health Care System, Temple, Texas
  - VA Medical Center, Hampton, Hampton, Virginia
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington
  - VA Medical Center, Clarksburg, Clarksburg, West Virginia
  - Wlliam S. Middleton Memorial Veterans Hospital, Madison, Madison, Wisconsin

REFERENCES:
- [Result] Wilt T. Expectant management or early intervention for clinically localized prostate cancer? What we need are randomized trials. Clinical Care For Prostatic Diseases. 1994 Jan 6; 1:1-9.
- [Result] Moon TD, Brawer MK, Wilt TJ. Prostate Intervention Versus Observation Trial (PIVOT): a randomized trial comparing radical prostatectomy with palliative expectant management for treatment of clinically localized prostate cancer. PIVOT Planning Committee. J Natl Cancer Inst Monogr. 1995;(19):69-71. No abstract available. PMID 7577210
- [Result] Wilt TJ, Brawer MK. Early intervention or expectant management for prostate cancer. The Prostate Cancer Intervention Versus Observation Trial (PIVOT): a randomized trial comparing radical prostatectomy with expectant management for the treatment of clinically localized prostate cancer. Semin Urol. 1995 May;13(2):130-6. No abstract available. PMID 7638470
- [Result] Wilt TJ, Brawer MK. The Prostate Cancer Intervention Versus Observation Trial (PIVOT). Oncology (Williston Park). 1997 Aug;11(8):1133-9; discussion 1139-40, 1143. PMID 9268976
- [Result] Wilt T. The importance of randomized treatment trials in early stage prostate cancer. New Developments in Prostate Cancer and Treatment. 1997 Feb 21; 2:29-35.
- [Result] Wilt TJ. Prostate cancer screening: practice what the evidence preaches. Am J Med. 1998 Jun;104(6):602-4. doi: 10.1016/s0002-9343(98)00127-2. No abstract available. PMID 9674725
- [Result] Wilt TJ. Uncertainty in prostate cancer care: the physician's role in clearing the confusion. JAMA. 2000 Jun 28;283(24):3258-60. doi: 10.1001/jama.283.24.3258. No abstract available. PMID 10866876
- [Result] Wilt TJ. Prostate carcinoma practice patterns: what do they tell us about the diagnosis, treatment, and outcomes of patients with prostate carcinoma? Cancer. 2000 Mar 15;88(6):1277-81. No abstract available. PMID 10717606
- [Result] Wilt T. Editorial comment. Urology. 2001 Nov 1; 58(6):964-965.
- [Result] Wilt TJ. Clarifying uncertainty regarding detection and treatment of early-stage prostate cancer. Semin Urol Oncol. 2002 Feb;20(1):10-7. doi: 10.1053/suro.2002.30393. PMID 11828353
- [Result] Wilt TJ. SPCG-4: a needed START to PIVOTal data to promote and protect evidence-based prostate cancer care. J Natl Cancer Inst. 2008 Aug 20;100(16):1123-5. doi: 10.1093/jnci/djn259. Epub 2008 Aug 11. No abstract available. PMID 18695131
- [Result] Kaplan SA, McConnell JD, Roehrborn CG, Meehan AG, Lee MW, Noble WR, Kusek JW, Nyberg LM Jr; Medical Therapy of Prostatic Symptoms (MTOPS) Research Group. Combination therapy with doxazosin and finasteride for benign prostatic hyperplasia in patients with lower urinary tract symptoms and a baseline total prostate volume of 25 ml or greater. J Urol. 2006 Jan;175(1):217-20; discussion 220-1. doi: 10.1016/S0022-5347(05)00041-8. PMID 16406915
- [Result] Wilt TJ, Brawer MK, Jones KM, Barry MJ, Aronson WJ, Fox S, Gingrich JR, Wei JT, Gilhooly P, Grob BM, Nsouli I, Iyer P, Cartagena R, Snider G, Roehrborn C, Sharifi R, Blank W, Pandya P, Andriole GL, Culkin D, Wheeler T; Prostate Cancer Intervention versus Observation Trial (PIVOT) Study Group. Radical prostatectomy versus observation for localized prostate cancer. N Engl J Med. 2012 Jul 19;367(3):203-13. doi: 10.1056/NEJMoa1113162. PMID 22808955
- [Result] Wilt TJ. Implications of the prostate intervention versus observation trial (PIVOT). Asian J Androl. 2012 Nov;14(6):815. doi: 10.1038/aja.2012.103. Epub 2012 Sep 17. No abstract available. PMID 22983306
- [Result] Wilt TJ. The Prostate Cancer Intervention Versus Observation Trial: VA/NCI/AHRQ Cooperative Studies Program #407 (PIVOT): design and baseline results of a randomized controlled trial comparing radical prostatectomy with watchful waiting for men with clinically localized prostate cancer. J Natl Cancer Inst Monogr. 2012 Dec;2012(45):184-90. doi: 10.1093/jncimonographs/lgs041. PMID 23271771
- [Result] Barry MJ, Andriole GL, Culkin DJ, Fox SH, Jones KM, Carlyle MH, Wilt TJ. Ascertaining cause of death among men in the prostate cancer intervention versus observation trial. Clin Trials. 2013;10(6):907-14. doi: 10.1177/1740774513498008. Epub 2013 Aug 29. PMID 23988464
- [Result] Wilt TJ, Scardino PT, Carlsson SV, Basch E. Prostate-specific antigen screening in prostate cancer: perspectives on the evidence. J Natl Cancer Inst. 2014 Mar;106(3):dju010. doi: 10.1093/jnci/dju010. Epub 2014 Mar 4. No abstract available. PMID 24594482
- [Derived] Wilt TJ, Vo TN, Langsetmo L, Dahm P, Wheeler T, Aronson WJ, Cooperberg MR, Taylor BC, Brawer MK. Radical Prostatectomy or Observation for Clinically Localized Prostate Cancer: Extended Follow-up of the Prostate Cancer Intervention Versus Observation Trial (PIVOT). Eur Urol. 2020 Jun;77(6):713-724. doi: 10.1016/j.eururo.2020.02.009. Epub 2020 Feb 21. PMID 32089359
- [Derived] Wilt TJ, Jones KM, Barry MJ, Andriole GL, Culkin D, Wheeler T, Aronson WJ, Brawer MK. Follow-up of Prostatectomy versus Observation for Early Prostate Cancer. N Engl J Med. 2017 Jul 13;377(2):132-142. doi: 10.1056/NEJMoa1615869. PMID 28700844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment begain in November 1994 and ended in January 2002 with follow-up through January 2010. We recruited men from 44 Department of Veterans Affairs sites and 8 National Cancer Institute sites.
Pre-assignment Details: A total of 13,022 men were entered into study logs as potentially eligible. Based upon further chart review, 6707 met age, comorbidity and prostate cancer specific criteria and received detailed information about the study. From these, 5023 were considered likely to be eligible and a total of 731 men agreed to participate.
Period: Overall Study
Arm/Group | Radical Prostatectomy | Watchful Waiting
Started | 364 | 367
Completed | 364 | 367
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radical Prostatectomy | Watchful Waiting | Total
Number analyzed (Participants) | 364 | 367 | 731
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 122 | 131 | 253
  >=65 years | 242 | 236 | 478
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (5.2) | 66.8 (5.6) | 66.9 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 364 | 367 | 731
Region of Enrollment [Number; unit: participants]
  United States | 364 | 367 | 731

OUTCOME MEASURES:

1. Primary Outcome: All Cause Mortality
Description: Number of deaths from any cause.
Time Frame: From date of randomization until date of death from any cause, assessed until end of study, up to 16 years
Measure: Count of Participants; unit: Participants
Arm/Group | Radical Prostatectomy | Watchful Waiting
Number analyzed (Participants) | 364 | 367
Participants | 171 | 183

ADVERSE EVENTS:
Arm/Group | Radical Prostatectomy | Watchful Waiting
Serious Adverse Events (participants affected / at risk) | 171/364 | 183/367
Other Adverse Events (participants affected / at risk) | 0/364 | 0/367
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radical Prostatectomy (N=364) | Watchful Waiting (N=367)
Death (General disorders) | 171 (171) | 183 (183)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes